CLINICAL TRIAL: NCT05355025
Title: WiserAD: A Randomised Trial of a Structured Online Intervention to Promote and Support Antidepressant Deprescribing in Primary Care.
Brief Title: WiserAD: The Effect of a Structured Online Intervention on Antidepressant Deprescribing in Primary Care
Acronym: WiserAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT19003; STOPS: A randomised trial of a (Other: University of Melbourne); GNT 1157337 (Other Grant/Funding Number: National Health and Medical Research Council)
Record Dates: First submitted 2022-03-30; First posted 2022-05-02 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Depression
Keywords: Deprescribing; Antidepressant; Tapering; Primary Care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Single blind, parallel-arm, randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomisation system will generate an email containing details of arm allocation which will be sent to the trial manager. The rest of the research team who will be blind to randomisation will only receive an email stating that a participant has been randomised. The treatment to which a participant is assigned will be determined by a computer generated pseudo-random code using random permuted blocks of varying size, created by the web developers and held on a secure server. Participants will be allocated with equal probability to each treatment arm and stratified by site (GP practice). Only the trial coordinator, or their nominee, will have password access to the randomisation data. Participants will not be blind to treatment group.
  Arm allocation will remain concealed to the research team until recruitment and follow up are complete. The trial coordinator will not be blind to allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be provided with a personal login code for the study web portal via automated email and encouraged to complete the initial components of the intervention which seek to determine participants' current support and management strategies and help them to understand their specific antidepressants. They will then complete the third component which contains three sub-sections to assist in creating a personal plan to help them cease their ADs: i) Management strategies for withdrawal symptoms and opportunities to discuss the plan with their GP or trusted Mental health worker; ii) Selecting a start time to begin tapering; iii) Print out of the personalised action plan to keep and share with supportive family and/or friends. Participants will also be required to complete a daily check-in through the portal which will check current symptoms and highlight any negative changes in emotional wellbeing, they will also receive texts reminders to complete these tasks.
  Interventions: Behavioral: WiserAD
- Usual care - Attention Control (Experimental): Participants allocated to the treatment as usual group will receive usual care plus attention control which comprises a link to the AD factsheet within the BeyondBlue website. This provides education material relevant to the participants' enrolment in the study but they will not be advised to cease or continue with their medication. GPs will not be advised of the participants allocated to this treatment arm.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: WiserAD — See "Arms"
  Arms: Intervention
Behavioral: Attention control — See "Arms"
  Arms: Usual care - Attention Control

SUMMARY:
The use of antidepressants (ADs) is increasing globally, including within Australia, which has one of the highest rates of AD prescribing. Despite clear benefits for many people, there is reason to believe that the ongoing use of these medications is often not properly monitored or stopped (deprescribed) when a person returns to better Mental health. This trial sets out to test how well an online support tool (WiserAD) can help patients and their general practitioner to manage the careful and appropriate reducing and stopping of antidepressants, in primary care patients.

DETAILED DESCRIPTION:
Antidepressants (ADs) have significantly improved the health and wellbeing for very many people and their success in enabling those with depression to retain their quality of life has undoubtedly led to their widespread use around the globe. However, the success of ADs has also led to a significant and unnecessary clinical and economic burden on the healthcare system and patients, through over prescribing, most often in cases when they are no longer of therapeutic use.

Such inappropriate medicine use (defined as use that is going against clinical guidelines) is a significant financial and clinical challenge for healthcare providers globally. Recent figures show that alongside the US, UK and parts of Northern Europe, Australia now has one of the world's highest AD prescribing rates with a total cost of over $200 million per year. In 2015-2016 alone there were more AD prescriptions than people: 24.72 million - up 20% since 2012. Significantly, much of this this is due to an excess of long term users rather than an increase in the number of people being newly diagnosed with major depressive disorder (MDD) or other disorders for which ADs are prescribed (e.g. anxiety). In a recent study by this group a cohort of almost 800 primary care patients with depressive symptoms showed that only 15% of long term users satisfied clinical criteria for long term AD use. There is relatively little research that explores the long term effects of AD use but there are indications that it can be harmful. In many cases, long term use can be linked to a range of severe side effects including increased risk of cardiovascular events, gastrointestinal bleeding and diabetes.

Psychological dependence is another problem facing users and stems from a perceived need to take ADs for fear of a relapse. That fear, shared by doctors, explains why AD use is unnecessarily protracted, even though it may undermine patients' autonomy and resilience, becoming less likely to self-manage or willing to stop their AD medication. Crucially, the evidence for relapse comes primarily from studies on AD users for whom guidelines recommend continued treatment (those who meet diagnostic criteria for moderate to severe major depressive disorder and have been receiving AD treatment for less than 12 months). In those with milder symptoms epidemiological research suggests that long-term AD use does not increase the likelihood of relapse and that that inappropriate long-term AD users can safely cease their medication. These findings are supported by a randomised controlled trial of AD cessation for primary care patients without current depression which showed a much smaller difference in relapse than previously thought.

Limiting AD use only to cases in which it is clinically indicated is in line with quality prescribing and will help to reduce costs and associated adverse events as well as the potential benefit of improving long-term mental health outcomes for patients. Although they are not addictive research has shown that ADs are more difficult to cease than other medications and previous studies have demonstrated limited success in deprescribing trials of antidepressants compared to other medications suggesting that a more intensive, patient-focused intervention is required to support successful de-prescribing. The WiserAD study will test whether a novel, structured approach to deprescribing antidepressants is more effective than usual practice in enabling GPs to help patients cease (or decrease) their AD medication whilst maintaining their mental health and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* Stable on AD for >=12m (no depressive episodes)
* No history of recurrent depression
* Sufficient English language proficiency to provide informed consent
* No or mild depressive symptoms (PHQ-9)
* Low risk of Suicide or Self-harm
* Agree to consider reviewing their AD use
* Agree to be randomized into the study
* Willing to provide informed consent

Exclusion Criteria:

* Moderate/severe depressive symptoms (PHQ-9 ≥10) at study entry or history of severe or recurrent depression
* Experienced a major life event in the past 3 months, or foresee one occurring in the next 3 months (e.g. trauma, grief, loss of role, major health issue, financial crisis)
* Continued AD use indicated for other condition (e.g. anxiety)
* Currently prescribed a non-SSRI/SNRI AD, antipsychotic, or mood stabiliser
* No internet access.

Exclusion Criteria:

Those currently experiencing a major life event in the next 3 months Currently using ADs for any other health condition (other than depression) Currently using non-SSRI or SNRI ADs, antipsychotics, or other mood stabiliser medication Have no daily access to the internet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-08-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients successfully ceasing ADs at 6-months post baseline | Primary outcome is at 6-months post baseline.
  Successful cessation is defined as no AD use and the absence of clinically significant depressive symptoms

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline, 3-, 6-, 12-, 18- and 24-months.
  9-items, 4-point likert scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-27 with higher scores indicating higher levels of depressive symptoms.
General Anxiety Disorder-7 (GAD-7) | Baseline, 3-, 6-, 12-, 18- and 24-months.
  7-items, 4-point likert scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-21 with higher scores indicating higher levels of anxiety.
Patient Activation Measure (PAM) | Baseline, 3-, 6-months.
  13-item measure that assesses patient knowledge, skill, and confidence for self-management. 4-point likert scale ranging from 1 (disagree strongly) to 4 (agree strongly) plus a "not applicable" option. Total PAM score is the raw score is divided by the number of items answered (excepting non-applicable items) and multiplied by 13. Then, this score is transformed to a scale with a theoretical range 0-100.
Assessment of Quality of Life (AQoL-4D) | Baseline, 3-, 6-, 12-, 18- and 24-months.
  12-item, likert scale (options differ depending on question). Scoring is for 4 dimensions (Independent Living, Mental Health, Relationships, Senses)
Resource Use Questionnaire (RUQ) | Baseline, 3-, 6-, 12-, 18- and 24-months.
  Study specific questionnaire measuring health resource use (e.g. doctor visits, medications taken).
Signs and Symptoms | 3-, 6-months.
  Study specific questionnaire asking about common AD side effects. Participants can enter up to 3 text response answers about any effects they have experienced.
Beliefs About Medication Questionnaire (BMQ) Antidepressant version | Baseline, 3-months.
  18-items, 5-point likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Scored across four domains (Specific Beliefs about Antidepressants - Necessity, Specific Beliefs about Antidepressants - Concerns, General beliefs about medicine - Overuse, General beliefs about medicine - Harms).
User Engagement Scale-Short Form (UES-SF) | 3- and 6-months.
  12-items, 5-point likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). An overall engagement score can be calculated by adding all of the items together and dividing by twelve.
Accountability Measurement Tool (AMT) | 3- and 6-months.
  12-items, 5-point likert scale ranging from 1 (Strongly disagree) to 5 (Strongly agree).
Medical Benefit Scheme (MBS) and the Pharmaceutical Benefit Scheme (PBS) data | Provided at completion of the study (patient data collected for duration of time in study - up to 2 years).
  Government collected data re: prescriptions and health service use for the duration of time in the study.
Proportion of patients successfully ceasing ADs at 6-months post baseline | Measured at 3-, 12-, 18-months to track deprescribing adherence.
  Successful cessation is defined as no AD use and the absence of clinically significant depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Gunn, PhD, Principal Investigator — University of Melbourne
Locations (1):
- Social Media, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No
IPD will not be available publicly due to confidential information being collected as part of the trial. Data collected as part of the trial will be for research purposes only.

REFERENCES:
- [Derived] Coe A, Gunn J, Allnutt Z, Kaylor-Hughes C. Understanding Australian general practice patients' decisions to deprescribe antidepressants in the WiserAD trial: a realist informed approach. BMJ Open. 2024 Feb 13;14(2):e078179. doi: 10.1136/bmjopen-2023-078179. PMID 38355180